CLINICAL TRIAL: NCT05195580
Title: Pre-pilot Study of Spine Registration Using 3D Scanning
Brief Title: Spine Registration Using 3D Scanning
Status: Terminated | Type: Observational
Why Stopped: Low enrollment of subjects
Sponsor: Advanced Scanners Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 01500
Record Dates: First submitted 2021-10-07; First posted 2022-01-19 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Spinal Fusion; Spinal Stenosis; Scoliosis; Spondylolisthesis
MeSH Terms: conditions — Spinal Stenosis; Scoliosis; Spondylolisthesis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Optical 3D Scanner — An optical 3D scanner used to register spine anatomy to surgical computer navigation systems.

SUMMARY:
The primary objective is to assess the capability of the device as measured by its consistency, its accuracy, and feedback from surgical staff over the study period.

ELIGIBILITY:
Inclusion Criteria:

1. Patients that require exposure of bony posterior spine anatomy for localization as standard of care.
2. Clinically planned for spine surgery.
3. Able to provide written informed consent from subject or subject's legal representative, using IRB approved consent form, and ability for subject to comply with the protocol requirements of the study.

Exclusion Criteria:

1. Language problems that would prevent from properly understanding instructions.
2. Requirement of an interpreter.
3. Patients who are excluded from consideration for the surgical procedure are therefore excluded from the research study.
4. Special populations: pregnant women, prisoners.
5. Minimally invasive spine surgery that does not expose the necessary bone/s.
6. Spine surgery without posterior exposure.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Subjects will be invited to participate from the Principal Investigator's clinic population. All subjects will be identified as requiring a spine surgery that meets the eligibility requirements.
Sampling Method: Non-Probability Sample
Enrollment: 2 (Actual)
Dates: Start 2021-08-31 (Actual); Primary Completion 2021-11-02 (Actual); Study Completion 2021-11-02 (Actual)

PRIMARY OUTCOMES:
Spine Registration | Throughout the surgical procedure
  Closely match the Advanced Scanners optical scan of the partially exposed surface of the patient vertebra to the corresponding patient's preoperative MRI and/or CT scan, thereby learning the position of the rest of the vertebra. This endpoint includes registration of the relevant preoperative MRI or CT scan portion to the portion scanned by Advanced Scanners.

SECONDARY OUTCOMES:
Vertebral Shift Measurement | Throughout the surgical procedure
  Use the intraoperative x-ray (typically O-arm) measurements taken at various times in the procedure to validate the capability of our scanner to determine relative shifts between vertebra as a function of time.
Determination Of Bony Exposure Requirements | Throughout the surgical procedure
  Measure the area of the exposed vertebra of registered adjacent segments. Bone regions will be identified in the scan mesh, segmented from the rest of the scan, and their areas determined directly from that surface region by integrating the area of the relevant mesh faces, in units of square millimeters or square centimeters.

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Bernstein, PhD, Study Director — Advanced Scanners Inc.
Locations (1):
- St. David's Round Rock Medical Center, Round Rock, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided
If data is shared, it will be anonymized.

REFERENCES:
- [Background] Arlt F, Chalopin C, Muns A, Meixensberger J, Lindner D. Intraoperative 3D contrast-enhanced ultrasound (CEUS): a prospective study of 50 patients with brain tumours. Acta Neurochir (Wien). 2016 Apr;158(4):685-694. doi: 10.1007/s00701-016-2738-z. Epub 2016 Feb 16. PMID 26883549
- [Background] Daanen, H. A. M. & Ter Haar, F. B. 3D whole body scanners revisited. Displays 34, 270-275 (2013).
- [Background] Hameeteman M, Verhulst AC, Vreeken RD, Maal TJ, Ulrich DJ. 3D stereophotogrammetry in upper-extremity lymphedema: An accurate diagnostic method. J Plast Reconstr Aesthet Surg. 2016 Feb;69(2):241-7. doi: 10.1016/j.bjps.2015.10.011. Epub 2015 Oct 22. PMID 26590631
- [Background] Kovacs L, Zimmermann A, Brockmann G, Guhring M, Baurecht H, Papadopulos NA, Schwenzer-Zimmerer K, Sader R, Biemer E, Zeilhofer HF. Three-dimensional recording of the human face with a 3D laser scanner. J Plast Reconstr Aesthet Surg. 2006;59(11):1193-202. doi: 10.1016/j.bjps.2005.10.025. Epub 2006 Mar 9. PMID 17046629
- [Background] Park HK, Chung JW, Kho HS. Use of hand-held laser scanning in the assessment of craniometry. Forensic Sci Int. 2006 Jul 13;160(2-3):200-6. doi: 10.1016/j.forsciint.2005.10.007. Epub 2005 Nov 9. PMID 16289612
- [Background] Zhang, D., Lu, G., Li, W., Zhang, L. & Luo, N. Palmprint Recognition Using 3-D Information. IEEE Transactions on Systems, Man, and Cybernetics, Part C (Applications and Reviews) 39, 505-519 (2009).